CLINICAL TRIAL: NCT01076244
Title: Single - Center, Prospective, Patient Outcomes Assessment of Minimally Invasive Lumbar Decompression With the Mild Devices in Patients With Symptomatic Central Canal Stenosis.
Brief Title: Vertos Mild - Post Market Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Pain Relief, Inc. (Other)
Collaborators: Vertos Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #D1; NCT01130350 (obsolete NCT alias)
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-02

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Minimally invasive lumbar decompression (Other)
  Interventions: Procedure: Minimally Invasive Lumbar Decompression

INTERVENTIONS:
Procedure: Minimally Invasive Lumbar Decompression — This minimally invasive procedure is performed under fluoroscopic image guidance through a dorsal approach to the spine. The patient is given local anesthesia and a sedative but needs to be responsive to the surgeon's questions for neurological monitoring. Under image guidance, the mild tools are inserted and positioned on the posterior spinal lamina, to the left or right of the spinous process. The tools are used to cut and remove tissue and bone from the posterior side of the lumbar spine to create a space inside the spine that can help decompress some of the spinal nerves.

SUMMARY:
This is a single-center study evaluating the outcomes of patients with painful lumbar spinal stenosis who were treated with the mild procedure (minimally invasive lumbar decompression. The patients will be followed for 6 months after the procedure.

DETAILED DESCRIPTION:
Approximately 50 patients at a single center will be enrolled and followed for a period of up to 26 weeks. Adult patients with symptomatic lumbar spinal stenosis who meet the enrollment criteria will be offered the mild procedure as an alternative to surgery or continued standard non-surgical medical management.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic and lumbar spinal stenosis caused by dorsal element hypertrophy
* Prior failure of conservative therapy and Oswestry Disability Index (ODI) >20%
* Radiologic evidence of lumbar spinal stenosis, ligamentum flavum hypertrophy (typically >2.5mm),confirmed by pre-op MRI/CT report
* Central canal cross sectional area clearly reduced per MRI/CT report
* If present, anterior listhesis < or = to 5.0mm (preferred) and deemed stable by the Investigator
* Able to walk at least 10 feet unaided before being limited by pain
* Available to complete 26 weeks of follow up
* A signed Consent Form is obtained from the patient
* Adults 18 years of age or older

Exclusion Criteria:

* Prior surgery at the intended treatment level
* Compound fracture with intraspinal retropulsion contributing to spinal stenosis
* Disabling back or leg pain from causes other than lumbar spinal stenosis
* Disc protrusion or osteophyte formation severe enough to confound study outcome
* Facet hypertrophy severe enough to confound study outcome
* Bleeding disorders and/or current use of anti-coagulants
* Use of acetylsalicylic acid (ASA) and/or non-steroidal anti-inflammatory drug (NSAID) within 5 days of treatment
* Epidural steroids with 3 weeks prior to procedure
* Inability of patient to lie prone for any reason with anesthesia support
* Metabolic wound healing pathologies that may be deemed by the Investigator to compromise the study outcomes
* Dementia and/or inability to give informed consent
* Pregnant and/or breastfeeding
* On workman's Compensation or considering litigation associated with back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Deer, MD, Principal Investigator — Center for Pain Relief, Inc
Locations (2):
- United States (2):
  - The Center for Pain Relief, Inc., Charleston, West Virginia
  - The Center for Pain Relief, Inc, Charleston, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled through one site (Center for Pain Relief) between March 2010 to January 2011.
Groups:
- Minimally Invasive Lumbar Decompression: Lumbar spinal stenosis patients exhibiting neurogenic claudication with predominance of ligamentum flavum hypertrophy were treated percutaneously using the mild Device Kit to decompress the target area.
Period: Overall Study
Arm/Group | Minimally Invasive Lumbar Decompression
Started | 46
Completed | 42
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Minimally Invasive Lumbar Decompression
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 66.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Secondary Outcome: Improvement in Functional Mobility
Description: Measured subjectively by the Oswestry Disability Index. Extent of disturbance in activities of daily living is subjectively reported using this validated instrument.Higher score indicate greater limitations in activity. The questionnaire is divided into 10 topics including pain intensity, personal care, lifting walking standing sitting, sleeping social life, traveling, employment/homemaking. Each topic is rated zero (no pain or no limitation) to 5 (high pain or very limited physically) based on typical pain and/or physical limitations. The worst possible score is 50 (100% disability) and the best score is zero (0% disability).Change from baseline to month 6 is reported below, where a positive value represents the baseline value minus the month 6 value.
Time Frame: baseline and month 6
Population: All available patients at six months were analyzed.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Minimally Invasive Lumbar Decompression
Number analyzed (Participants) | 42
units on a scale | 13.43 [8.42 to 18.43]
Statistical Analysis 1: Comparison: Minimally Invasive Lumbar Decompression; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; change from baseline = 13.43, 95% CI 2-sided [8.42 to 18.43], Standard Deviation 16.55

2. Secondary Outcome: Quality of Life as Measured by the Symptom Severity Scale of the Zurich Claudication Questionnaire (ZCQ).
Description: As a validated patient outcome tool specific to lumbar spinal stenosis, Zurich Claudication Questionnaire (ZCQ) captures symptom severity as a quality of life indicator. A mean score of 1 is the best possible outcome representing 'no pain' in symptom severity, whereas higher mean scores up to a maximum of 5 indicate worse patient symptoms. The symptom severity outcomes are presented below as change from baseline to month 6 where a positive value represents the baseline value minus the 6 month value. Treatment is considered 'successful' or 'clinically relevant' if the patient population has at least a 0.5 improvement in symptom severity.
Time Frame: Baseline and month 6
Population: All patients having a month six report report were analyzed.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Minimally Invasive Lumbar Decompression
Number analyzed (Participants) | 42
units on a scale | 1.07 [0.83 to 1.31]

3. Primary Outcome: Pain as Measured by Visual Analog Scale (VAS).
Description: A validated ten point scale was used where ten is the worst possible pain and zero represents complete lack of pain. The change from baseline to six months is presented below, where a positive value represents the baseline value minus the 6 month value.
Time Frame: Baseline and six months
Population: all available patients reporting at Month 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Minimally Invasive Lumbar Decompression
Number analyzed (Participants) | 42
units on a scale | 2.17 [1.17 to 3.16]
Statistical Analysis 1: Comparison: Minimally Invasive Lumbar Decompression; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; change from baseline = 2.17, 95% CI 2-sided [1.17 to 3.16], Standard Deviation 3.29

4. Secondary Outcome: Quality of Life as Measured by Physical Function Scale of the Zurich Claudication Questionnaire (ZCQ).
Description: For this ZCQ domain, a mean score of 1 is the best possible outcome representing 'no limitation' in physical function, whereas a mean score of 4 indicates worst physical function. Zurich Claudication physical function scale from this validated lumbar spine-specific measurement questionnaire are reported below as change from baseline to month 6. A positive value represents the baseline value minus the 6 month value. Treatment is considered clinically relevant when at least a 0.5 improvement is achieved.
Time Frame: Baseline and month 6
Population: All available patients at the month 6 reporting period were analyzed.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Minimally Invasive Lumbar Decompression
Number analyzed (Participants) | 42
units on a scale | 0.59 [0.34 to 0.84]

ADVERSE EVENTS:
Time Frame: Continuous from enrollment through follow-up period.
Arm/Group | Minimally Invasive Lumbar Decompression
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No